CLINICAL TRIAL: NCT00289614
Title: Patients With Renal Impairment and Diabetes Undergoing Computed Tomography
Brief Title: Patients With Renal Impairment and Diabetes Undergoing Computed Tomography (CT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: IOP 105
Record Dates: First submitted 2006-02-08; First posted 2006-02-10 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2008-01

CONDITIONS: Kidney Diseases
Keywords: contrast induced nephropathy
MeSH Terms: conditions — Kidney Diseases

INTERVENTIONS:
Drug: Iopamidol 370 mgI/dL

SUMMARY:
The main purpose of this study is to compare the incidence of contrast induced nephrotoxicity following the administration of Isovue (iopamidol) or Visipaque in diabetic patients with moderate to severe chronic renal impairment undergoing clinically indicated contrast enhanced multidetector computed tomography (MDCT). Serum creatinine will be measured before and up to 48-72 hours post dose.

ELIGIBILITY:
Inclusion Criteria:

* Referred for contrast enhanced MDCT
* Documented predose eGFR of greater than or equal to 20 and less than 60 mL/min/1.73m2
* Diagnosed as having diabetes mellitus

Exclusion Criteria:

* Unstable renal function
* Unstable diabetes
* Concurrent administration of nephrotoxic drugs
* Undergoing dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2006-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Increase in serum creatinine (SCr) at 48-72 hours post dose

SECONDARY OUTCOMES:
Decrease in estimated glomerular filtration rate (eGFR) at 48-72 hours post dose; occurrence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen S Bensel, CNMT, Study Director — Bracco Diagnostics, Inc
Locations (1):
- Bracco Diagnostics, Inc., Princeton, New Jersey, United States